CLINICAL TRIAL: NCT04618328
Title: A Study of All-trans Retinoic Acid in the Treatment of Immune Thrombocytopenia
Brief Title: A Study of ATRA in the Treatment of ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Beijing Hospital (Other Government); Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5000 offer
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: ATRA is used to treat ITP patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATRA treatment group (Experimental): ATRA is given at a daily dose of 10 mg twice daily orally for 12 weeks
  Interventions: Drug: all trans retinoic acid

INTERVENTIONS:
Drug: all trans retinoic acid — ATRA is given concomitantly at a daily dose of 10 mg twice daily orally for 12 weeks
  Other Names: ATRA

SUMMARY:
An open-label, multicenter study to compare the efficacy and safety of ATRA for the treatment of adults with primary immune thrombocytopenia (ITP)

DETAILED DESCRIPTION:
The investigators are undertaking an open-label, single-arm, multicenter trial of adults patients with ITP in China. Patients with treatmant naive ITP were given ATRA treatment. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed newly-diagnosed, treatment-naive ITP;
2. Platelet counts <30×109/L ;
3. Platelet counts < 50×109/L and significant bleeding symptoms (WHO bleeding scale 2 or above);
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit;
2. Received first-line and second-line ITP-specific treatments (eg, steriods, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit;
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study.
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections;
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia);
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period;
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
8. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 6 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up

SECONDARY OUTCOMES:
complete response (CR) | day 14
  complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding.
Response (R) | day 14
  Response (R) as platelet count more than 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.
Number of patients with bleeding | 6 months
  Number of patients with bleeding complication ( WHO bleeding score).
Number of patients with adverse events | 6 months
  Number of patients with adverse events
Time to response | 6 months
  The time from starting treatment to time of achievement of CR or R
Duration of response (DOR) | 6 months
  Duration of response at 6-month follow up.
loss of response | 6 months
  Platelet counts below 100 x 109/L or bleeding (from CR) or platelet counts below 30 x 109/L, less than 2-fold increase of baseline platelet count or bleeding (from R)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, Doctor, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China